CLINICAL TRIAL: NCT04784871
Title: Promoting Wellbeing: A Randomized Controlled Trial of the Five Ways to All Intervention
Brief Title: Promoting Wellbeing: The Five Ways to All Intervention
Acronym: 5WaysA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Norwegian Institute of Public Health (Other Government); Norwegian Council for Mental Health (Other); The Dam Foundation (Other)
Responsible Party: Principal Investigator, Monica Beer Prydz, Principal Investigator, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 461814
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Wellbeing; Health Attitude; Quality of Life
Keywords: Wellbeing; Health promotion; Web-based intervention

STUDY DESIGN:
Intervention Model Description: The design is a randomized controlled trial (RCT) with one intervention group and two wait-list control groups. The goal with this design is to demonstrate the initial efficacy and feasibility of the 5WaysA intervention. We have one active control group writing activity log and one inactive not getting any tasks while waiting. The effect analysis will involve a comparison of self-reported wellbeing at different measurement points, using a two-way mixed measures ANOVA. In addition, PI will run a longitudinal analysis using linear mixed (multilevel) models on the data from all 5-6 measurement time points. Mixed modelling is a flexible way to handle unbalanced data in case of non-registration and repeated observations. The models allow PI to investigate the effects of the intervention and test the hypotheses of group and individual development in wellbeing while controlling for both stable and time-varying covariates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 5waysA Intervention (Experimental): The intervention, 5WaysA, is a 10 week modified web-based version of the original Five Ways to Wellbeing course. The intervention consists of a two-hour main webinar with live lecturing from a facilitator introducing the Five Ways to Wellbeing framework and teaching the participants how to implement the five health promotive activities in life, a booster session webinar four weeks later, as well as an SMS message twice a week in the six following weeks. Each SMS encourages participants to engage in one of the five activities, register activities/goals and queries about the degree of participation in the activity introduced in the previous SMS.
  Interventions: Behavioral: 5waysA Intervention
- 5waysA Active wait-list control (Other): The active wait-list control group will get the same intervention as the interventions group, five months later. The active wait-list control group will be encouraged (in SMS messages) to write down an activity log once a week in ten weeks, while waiting. The participants in this group will also answer questionnaires after the intervention group has finished the intervention
  Interventions: Behavioral: 5waysA Active wait-list control
- 5waysA Inactive wait-list control (Other): The inactive wait-list control group will get the same intervention as the interventions group, five months later. The inactive wait-list control group will not do anything specific while waiting for the intervention. The participants in this group will also answer questionnaires after the intervention group has finished the intervention
  Interventions: Behavioral: 5waysA Inactive wait-list control

INTERVENTIONS:
Behavioral: 5waysA Intervention — Web-based 10 week intervention, encouraging participants engaging in five potential health promoting activities: 1. Be active, 2. Take notice, 3. Keep learning, 4. Connect and 5. Give.
  Arms: 5waysA Intervention
Behavioral: 5waysA Active wait-list control — Writing activity log in the waiting time. Then, after five months and the writing of activity log, the participants get the web-based intervention and SMS massages, which encourage the participants to engage in five potential health promoting activities: 1. Be active, 2. Take notice, 3. Keep learning, 4. Connect and 5. Give.
  Arms: 5waysA Active wait-list control
Behavioral: 5waysA Inactive wait-list control — No activity while the participants wait. After five months of waiting, the participants get the web-based intervention and SMS messages, which encourage participants engage in five potential health promoting activities: 1. Be active, 2. Take notice, 3. Keep learning, 4. Connect and 5. Give.
  Arms: 5waysA Inactive wait-list control

SUMMARY:
This project is funded by Stiftelsen Dam and is a cooperation between The Norwegian Council for Mental Health (NCMH) and PROMENTA research group at the University of Oslo. Low-cost and evidence-based health promoting public health tools are urgently needed in Norwegian municipalities, to meet both current and future challenges with mental health and wellbeing. The aim in this randomized controlled trail is to test if a shorter, 10 week web-based version (The Five Ways to All, "5WaysA"), of an already established course (Five Ways to Wellbeing course), can promote wellbeing and mastery in the general population. The principal investigator will investigate to what extend the effects are short-term and long-term (i.e., 10 weeks, 18 weeks and 12 months after starting to receive the 5WaysA intervention).

DETAILED DESCRIPTION:
Background:

The need for effective, low-cost and evidence-based tools to prevent illness and promote health in the population is paramount. Norway, along with other countries in the Western world, is currently facing major health and welfare-related challenges. Demographic changes, lifestyle related diseases and work absence are threatening the sustainability of the Norwegian welfare state. Non-communicable diseases, including mental illness, currently account for 65% of the total disease burden in Norway and 50% of Norwegians are likely to meet diagnostic criteria for a mental disorder some time during their life span. Traditional treatment and care options tend to be costly and time consuming, and to depend on highly skilled specialist human resources. Systematic findings also indicate that population-based (i.e., universal, targeting the general population) measures often result in larger population health gains than selective and indicated measures targeting only those with excess risk. According to the paradox of prevention, when disease risk is common, universal interventions directed towards the whole population before illness occurs, are more effective than interventions targeting high risk groups after symptoms have emerged. The Covid-19 pandemic and associated social distancing measures have corroborated the need for digital solutions. Web-based interventions may reach a large number of participants, utilizing a very modest amount of both human and financial resources.

The aim:

This study aims to test a potentially effective low-cost health and wellbeing promotive web-based intervention targeting the general population in Norwegian municipalities. The intervention is based on the Five Ways to Wellbeing framework developed for British health authorities in 2008. This framework, and the intervention to be tested, provides participants with knowledge on simple, sustainable activities that may strengthen their subjective wellbeing (SWB), mastery, health and social relations, thereby also reducing the risk of common mental health problems such as depression and anxiety. The study will be conducted in close collaboration with municipal stakeholders and important user groups. Thus, the principal investigator (PI) will investigate effects of a low-cost health and wellbeing promotive public health tool based on the evidence-base of Five Ways to Wellbeing. To date, nobody has tested the Five Ways-concept in such a format. Proved effective, this web-based 5WaysA intervention, may have a significant impact on the public health of inhabitants in the municipalities.

Main hypothesis:

The web-based intervention 5WaysA will improve wellbeing and mastery and hence provide the municipalities with an effective measure for mental health promotion.

Research questions:

1. To what extent does participation in the web-based 5WaysA intervention lead to improved wellbeing, mental health and mastery in the general population?
2. To what extent are the effects short-term and long-term (i.e., 10 weeks, 18 weeks and 12 months after starting to receive the 5WaysA intervention)?
3. What mechanisms explain potential improvements in wellbeing?

   1. For whom is this intervention effective (i.e., is the effect moderated by e.g. gender, age, education)?
   2. What mechanisms (e.g., regular practicing of 5Ways actions, increased social activity or support) explain intervention effects?

Sample and recruitment:

The PI plan to recruit a minimum of 1500 participants from the general population in Norwegian municipalities. The participants will be randomized to either an intervention group (n=750), or to one of two wait-list control groups (active control, n=375) (inactive control, n =375). The wait-list control groups will receive the intervention three to five months later. The PI expect high drop-out (up to 50 %) since this has been the situation in other studies investigating online interventions in a general population. The PI is also unsure about how much time the municipalities have to help PI with the recruitment process, because of a high work load in the municipalities during the pandemic of Covid-19.

Note (June 19, 2021): PI was only able to recruit 226 participants in spring 2021. PI will continue the recruitment process and do another round of the intervention in fall 2021. This will not be registered as a new study, and is regarded as part of the current study

Procedures:

The web-based 10 week intervention consist of one main webinar (two hours at Zoom), a booster session webinar five weeks later and SMS messages twice a week in the the six following weeks. The webinars will be live lectures with an independent trained facilitator. The SMS messages will be sent out by the PI (via Nettskjema) to all participants while they are in the interventions period. Questionnaires will be administrated and distributed by the PI by using the Nettskjema and Services for sensitive data (TSD) tools. The measurements will also be conducted use of Nettskjema and TSD.

Power analysis:

The PI assume that we can recruit a minimum of 1500 participants, but high drop-out is expected. An a priori power analysis was conducted using G*Power3 to test the interaction effect in a mixed ANOVA, using a two-tailed test, assuming a small effect size (f = .10), and an alpha of .05. The assumed effect size (f=0.1) was chosen as it is of the same magnitude (lower bound) as has been reported by other universal interventions with wellbeing as the outcome measure. The result showed that if PI attained a total sample of 750 participants at the second measurement point (attrition of 50%), PI would have power of .999 to detect a group by time interaction. The high level of statistical power will enable PI to investigate both moderators and mediators of the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old

Exclusion Criteria:

* under 18 years old

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 970 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Wellbeing (Subjective wellbeing, global life satisfaction) | 12 months
  Satisfaction With Life Scale (Diener, 2009) Scoring: 31 - 35 Extremely satisfied, 26 - 30 Satisfied, 21 - 25 Slightly satisfied, 20 Neutral,15 - 19 Slightly dissatisfied, 10 - 14 Dissatisfied and 5 - 9 Extremely dissatisfied
Wellbeing (Psychological wellbeing, self-perceived success in different aspects of life) | 12 months
  Flourishing Scale (Diener et. al 2009). Scores from 8 (lowest possible wellbeing) to 56 (highest possible wellbeing).

SECONDARY OUTCOMES:
Mastery | 12 months
  Pearlin and Schooler (1978). Scores from 7-49, the higher score the higher mastery.
Mental health (symptoms of depression and anxiety,) | 12 months
  Hopkins Symptom Checklist-8 (HSCL-8). Scores from 0-32, the higher score the more symptoms (Tambs & Røysamb, 2014)
Social life | 12 months
  Oslo Social Support Scale-3 (OSS-3) Scores: 3-14, where high levels represent high levels of social support
Physical health | 12 months
  Two questions from 12-Item Short Form Survey (SF-12) Scores: 12-47, where higher scores mean poorer health

OTHER OUTCOMES:
Work participation | 12 months
  Single question
Five ways to wellbeing- activities: connect, keep learning, take notice and give. | 12 months
  Four questions with scores in a range from 0 to 10, the higher score the more engaged in the activity.
Five ways to wellbeing- activity: be active. Frequency, duration and intensity. | 12 months
  Three single questions from The Norwegian County Survey. Frequency; scores range from 0 to 6 (the higher score the more often physical active). Intensity; scores from 0-3 (the higher score the higher intensity). Duration: Scores from 0-4 (the higher score the longer duration)
Basic feelings | 12 months
  Questions about feelings (happy, sad, irritated, lonely, engaged, calm, curious/interested). Scores rage from 0 to 10. 0 indicating not having the feeling at all, 10 indicating experience the feeling a lot.
Optimistic about the future | 12 months
  On single question. Score from 0 to 10, the higher score the more optimistic

CONTACTS AND LOCATIONS:
Overall Officials: Monica B Prydz, Cand.psychol, Principal Investigator — University of Oslos
Locations (1):
- Monica Beer Prydz, Asker, Norge, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prydz MB, Czajkowski NO, Eilertsen M, Roysamb E, Nes RB. A Web-Based Intervention Using "Five Ways to Wellbeing" to Promote Well-Being and Mental Health: Randomized Controlled Trial. JMIR Ment Health. 2024 May 20;11:e49050. doi: 10.2196/49050. PMID 38767958

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT04784871/Prot_SAP_000.pdf